CLINICAL TRIAL: NCT05941871
Title: Diet and Chronotype: a Randomized Controlled Trial to Evaluate the Effects of a Chronotype-adapted Diet on Weight Loss in Overweight/Obese Subjects
Brief Title: Chronotype-adapted Diet and Weight Loss
Acronym: CHRONODIET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Francesco Sofi, Professor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRONODIET
Record Dates: First submitted 2023-05-18; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Overweight and Obesity
Keywords: Chrono-nutrition; Circadian rhythms; Chronotype; Weight loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Randomised and controlled trial with 2 arms of intervention
Masking Description: In this trial blinding of experimenters will not be possible as they will have to administer the chronotype diet in the intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Group that will follow a low-calorie diet with a standard daily energy distribution for 4 months
  Interventions: Other: Dietary intervention - control group
- Intervention (Experimental): Group following a low-calorie diet with a different daily energy distribution according to their chronotype for 4 months
  Interventions: Other: Dietary intervention - intervention group

INTERVENTIONS:
Other: Dietary intervention - intervention group — Low-calorie diet for 4 months with a different daily energy distribution according to the chronotype:
  * Morning chronotype: 50% of kcal administered before lunch and 15% in the second part of the day (specifically: 40% at breakfast, 10% in the morning snack, 35% at lunch, 5% at afternoon snack and 10% at dinner)
  * Evening chronotype: 15% of kcal given before lunch and 50% in the second half of the day (specifically: 10% of kcal at breakfast, 5% in the morning snack, 35% at lunch, 10% at snack time and 40% at dinner)
  Arms: Intervention
Other: Dietary intervention - control group — Group that will follow a low-calorie diet with a standard daily energy distribution (20% of kcal at breakfast, 10% in the morning snack, 35% at lunch, 10% at afternoon snack and 25% at dinner) for 4 months
  Arms: Control

SUMMARY:
In humans, prolonged alterations in the circadian rhythm have been linked to cognitive impairments, premature ageing, and oncological and metabolic disorders such as diabetes and obesity. Obesity, in particular, is an ever-increasing condition with innumerable deleterious effects on human health. In recent years, studies have shown a relationship between a person's chronotype (morning or evening) and eating habits, as well as the importance of adapting these habits to physiological rhythms. Furthermore, it has been suggested that customising the caloric distribution of meals according to personal circadian rhythms may influence body weight and be one of the strategies to control overweight and obesity. In spite of the strong interest in this topic and the increasing number of observational studies conducted, there is currently a lack of intervention studies evaluating whether a low-calorie diet that takes into account the individual chronotype may be more effective than a standard low-calorie diet in the treatment of overweight and/or obesity.

DETAILED DESCRIPTION:
Background

Society has changed enormously in recent decades and this has had a strong impact on the processes regulating circadian rhythms, in particular the sleep-wake and fasting-eating cycles. The 'normalisation' of the environment, favoured by technological progress, has in fact caused light pollution, noise pollution, excessive thermoregulation, continuous work shifts and disordered eating, leading to an uncoordinated circadian cycle with consequences on physical and mental balance. In humans, prolonged alterations of the biological clock have been linked to cognitive disorders, premature ageing, and oncological and metabolic diseases such as diabetes and obesity. Obesity, in particular, is a condition with innumerable negative effects on human health.

In recent years, a new branch of nutritional research has aroused growing interest in the scientific community: this is chrono-nutrition, which combines elements of nutritional research with elements of chronobiology and studies the impact of eating times on health. The first to use the term "chrono-dystrophy" as a chronic desynchronisation of circadian rhythms were Erren and colleagues, who in their work reported how a loss of synchronisation between environmental signals and physiological processes can lead to alterations in the communication between the central nervous system and peripheral clocks and a change in the subject's metabolism. Subsequently, numerous studies have evaluated the impact of the thirteen dimensions of eating behaviour - timing, frequency and regularity - on health, hypothesising a possible role of the individual circadian rhythm, or chronotype, on the risk of developing overweight and/or obesity. Recent data have demonstrated a relationship between a person's chronotype (morning or evening) and eating habits, as well as the importance of adapting these habits to physiological rhythms. Furthermore, it has been suggested that customising the caloric distribution of meals according to personal circadian rhythms may influence body weight and be one of the strategies to control overweight and obesity. Indeed, recent research has shown that calories ingested at different times of the day have different effects on energy utilisation, leading to differential weight loss, even in the presence of isocaloric quantities.

Despite the strong interest in this topic and the increasing number of observational studies conducted, there is currently a lack of intervention studies evaluating whether a dietary regimen can be used to control body weight. Evidence to date suggests that in order to increase the effectiveness of low-calorie diets, it may be of great interest to consider not only patients' daily energy expenditure but also their circadian preferences. Overall, chrono-nutrition could mediate the effects between sleep, diet and urbanisation, but further research is needed to elucidate the precise physiological and metabolic mechanisms underlying this phenomenon, the importance of chronotype for metabolic health and its impact on public health.

Objectives of the study

The objectives of the study are to compare the effects of a diet with a daily calorie distribution adapted to the individual chronotype with a control diet with a conventional daily calorie distribution. The primary outcome is weight change from baseline. Secondary outcomes are changes in body mass index (BMI), percentage of fat mass, biochemical parameters and gut microbiota profile.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese condition (BMI≥25 kg/m2)
* age between 18 and 65 years
* willing to give informes consent

Exclusion Criteria:

* chronic illnesses or unstable conditions (e.g. cancer, kidney or liver disease, inflammatory-intestinal disease, cognitive decline, psychiatric disease)
* drug therapies (use of corticosteroids, antidiabetic drugs)
* pregnancy or intention to become pregnant in the next 12 months
* breastfeeding
* current or recent (last 3 months) adoption of a low-calorie diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-03-06 (Estimated); Study Completion 2025-03-06 (Estimated)

PRIMARY OUTCOMES:
Weight change | 4 months
  Measurement of body weight change from baseline in kg

SECONDARY OUTCOMES:
Body mass index (BMI) changes | 4 months
  Measurement of BMI change from baseline. Weight and height will be combined to report BMI in kg/m^2
Fat mass changes | 4 months
  Measurement of fat mass change from baseline. Percentage of fat mass will be assessed using the Akern bioelectrical impedance analyser (model SE 101)
Fasting Blood Glucose changes | 4 months
  Measurement of blood glucose concentration change from baseline in mg/dL
Total cholesterol changes | 4 months
  Measurement of total cholesterol change from baseline in mg/dL
LDL-cholesterol changes | 4 months
  Measurement of LDL cholesterol change from baseline in mg/dL
HDL-cholesterol changes | 4 months
  Measurement of HDL cholesterol change from baseline in mg/dL
Triglycerides changes | 4 months
  Measurement of triglycerides change from baseline in mg/dL
Aspartate transaminase changes | 4 months
  Measurement of aspartate transaminase change from baseline in U/l
Alanine transaminase changes | 4 months
  Measurement of alanine transaminase change from baseline in U/L
Gamma gamma-glutamyl transferase changes | 4 months
  Measurement of gamma-glutamyl transferase change from baseline in U/L
Urea changes | 4 months
  Measurement of urea change from baseline in mg/dL
Creatinine changes | 4 months
  Measurement of creatinin change from baseline in mg/dL
Uric acid changes | 4 months
  Measurement of uric acid change from baseline in mg/dL
Gut microbiota changes | 4 months
  Measurement of gut microbiota profile change from baseline. Each subject will be asked for a stool sample at the start of the study and at the end after 4 months in order to analyse the composition of the gut microbiota and short-chain fatty acids production

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Sofi, MD, PhD, Study Director — Unit of Clinical Nutrition University Hospital of Careggi, Florence
Locations (1):
- Unit of Clinical Nutrition, University Hospital of Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Almoosawi S, Vingeliene S, Gachon F, Voortman T, Palla L, Johnston JD, Van Dam RM, Darimont C, Karagounis LG. Chronotype: Implications for Epidemiologic Studies on Chrono-Nutrition and Cardiometabolic Health. Adv Nutr. 2019 Jan 1;10(1):30-42. doi: 10.1093/advances/nmy070. PMID 30500869
- [Background] Erren TC, Reiter RJ. Defining chronodisruption. J Pineal Res. 2009 Apr;46(3):245-7. doi: 10.1111/j.1600-079X.2009.00665.x. Epub 2009 Feb 9. PMID 19215573
- [Background] Horne JA, Ostberg O. A self-assessment questionnaire to determine morningness-eveningness in human circadian rhythms. Int J Chronobiol. 1976;4(2):97-110. PMID 1027738
- [Background] Galindo Munoz JS, Gomez Gallego M, Diaz Soler I, Barbera Ortega MC, Martinez Caceres CM, Hernandez Morante JJ. Effect of a chronotype-adjusted diet on weight loss effectiveness: A randomized clinical trial. Clin Nutr. 2020 Apr;39(4):1041-1048. doi: 10.1016/j.clnu.2019.05.012. Epub 2019 May 21. PMID 31153674
- [Background] Lotti S, Pagliai G, Colombini B, Sofi F, Dinu M. Chronotype Differences in Energy Intake, Cardiometabolic Risk Parameters, Cancer, and Depression: A Systematic Review with Meta-Analysis of Observational Studies. Adv Nutr. 2022 Feb 1;13(1):269-281. doi: 10.1093/advances/nmab115. PMID 34549270
- [Background] Maukonen M, Kanerva N, Partonen T, Kronholm E, Konttinen H, Wennman H, Mannisto S. The associations between chronotype, a healthy diet and obesity. Chronobiol Int. 2016;33(8):972-81. doi: 10.1080/07420528.2016.1183022. Epub 2016 May 31. PMID 27246115
- [Background] Maukonen M, Kanerva N, Partonen T, Kronholm E, Tapanainen H, Kontto J, Mannisto S. Chronotype differences in timing of energy and macronutrient intakes: A population-based study in adults. Obesity (Silver Spring). 2017 Mar;25(3):608-615. doi: 10.1002/oby.21747. PMID 28229553
- [Background] Patterson F, Malone SK, Lozano A, Grandner MA, Hanlon AL. Smoking, Screen-Based Sedentary Behavior, and Diet Associated with Habitual Sleep Duration and Chronotype: Data from the UK Biobank. Ann Behav Med. 2016 Oct;50(5):715-726. doi: 10.1007/s12160-016-9797-5. PMID 27056396
- [Background] Potter GD, Skene DJ, Arendt J, Cade JE, Grant PJ, Hardie LJ. Circadian Rhythm and Sleep Disruption: Causes, Metabolic Consequences, and Countermeasures. Endocr Rev. 2016 Dec;37(6):584-608. doi: 10.1210/er.2016-1083. Epub 2016 Oct 20. PMID 27763782
- [Background] Roenneberg T, Merrow M. The Circadian Clock and Human Health. Curr Biol. 2016 May 23;26(10):R432-43. doi: 10.1016/j.cub.2016.04.011. PMID 27218855
- [Background] Ruddick-Collins LC, Johnston JD, Morgan PJ, Johnstone AM. The Big Breakfast Study: Chrono-nutrition influence on energy expenditure and bodyweight. Nutr Bull. 2018 Jun;43(2):174-183. doi: 10.1111/nbu.12323. Epub 2018 May 8. PMID 29861661
- [Background] Sofi F, Dinu M, Pagliai G, Cesari F, Marcucci R, Casini A. Mediterranean versus vegetarian diet for cardiovascular disease prevention (the CARDIVEG study): study protocol for a randomized controlled trial. Trials. 2016 May 4;17(1):233. doi: 10.1186/s13063-016-1353-x. PMID 27145958
- [Background] Sofi F, Dinu M, Pagliai G, Pierre F, Gueraud F, Bowman J, Gerard P, Longo V, Giovannelli L, Caderni G, de Filippo C. Fecal microbiome as determinant of the effect of diet on colorectal cancer risk: comparison of meat-based versus pesco-vegetarian diets (the MeaTIc study). Trials. 2019 Dec 9;20(1):688. doi: 10.1186/s13063-019-3801-x. PMID 31815647
- [Derived] Dinu M, Lotti S, Pagliai G, Napoletano A, Asensi MT, Giangrandi I, Marcucci R, Amedei A, Colombini B, Sofi F. Effects of a chronotype-adapted diet on weight loss, cardiometabolic health, and gut microbiota: study protocol for a randomized controlled trial. Trials. 2024 Feb 28;25(1):152. doi: 10.1186/s13063-024-07996-z. PMID 38419068